CLINICAL TRIAL: NCT02790164
Title: Continuous Neuromuscular Blocking Agent for out-of Hospital Cardiac Arrest; Multicenter Randomized Controlled Trial
Brief Title: Continuous NMB in PCAS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chun Song Youn (Other)
Collaborators: The Catholic University of Korea (Other); Uijeongbu St. Mary's Hospital (Unknown); Chonnam National University Hospital (Other); Asan Medical Center (Other); Hanil General Hospital (Unknown); Ulsan Universty Hospital (Unknown); Hanyang University Guri Hospitall (Unknown)
Responsible Party: Sponsor-Investigator, Chun Song Youn, Professor, Seoul St. Mary's Hospital
Organization: Seoul St. Mary's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5-2016-B0001-00003
Record Dates: First submitted 2016-05-25; First posted 2016-06-03 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Out-of-hospital Cardiac Arrest
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest | interventions — Rocuronium; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rocuronium (Experimental): Patients will receive a bolus dose of 0.6 mg/kg, then a continuous I.V. infusion of 0.3-0.6 mg/kg/hr as per standard intensive care unit practice.
  Interventions: Drug: Esmeron
- Usual Care (Placebo Comparator): Patients will receive 100 mL of normal saline over 5-10 minutes at the beginning of the study in addition to usual care.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Esmeron — Neuromuscular Blockade
  Other Names: Rocuronium
  Arms: Rocuronium
Drug: Saline — Normal Saline
  Arms: Usual Care

SUMMARY:
The main purpose of this study is to test the hypothesis that continuous NMB could improve outcome in cardiac arrest patients treated with therapeutic hypothermia.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (older than 19)
2. OHCA with sustained ROSC
3. Comatose (i.e., not following commands) following ROSC
4. Undergoing targeted temperature management (TTM)
5. Time of enrollment ≤ 6hrs from ROSC

Exclusion Criteria:

1. Pre-existing dementia, brain injury, or dependence on others for ADLs (CPC > 3)
2. Traumatic etiology for cardiac arrest
3. Protected population (pregnant, prisoner)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2016-05; Primary Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Lactate levels 24 hours after initiation of study drug | 24 hours

SECONDARY OUTCOMES:
Lactate change over time | 0, 12, 24, 36 hrs
Survival | Duration of hospitalization, limit 180 days
  in-hospital survival
Good neurological outcome | Duration of hospitalization, limit 180 days
  Modified Rankin Scale
Length of intensive care unit stay | Duration of ICU stay, limit 180 days

CONTACTS AND LOCATIONS:
Overall Officials: Chun Song Youn, MD, Principal Investigator — Seoul St. Mary's Hospital
Locations (1):
- Seoul St. Mary's Hospital, Seoul, Seoul, South Korea